CLINICAL TRIAL: NCT01202552
Title: Two-site Intradermal Influenza Vaccination in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Saovabha Memorial Institute (Other)
Responsible Party: Principal Investigator, Suda Sibunruang, Principal investigator, Queen Saovabha Memorial Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TIC 5301
Record Dates: First submitted 2010-09-13; First posted 2010-09-16 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Influenza
Keywords: influenza; aged; intradermal injection
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- group 1 (Experimental): receives a single intramuscular dose of 0.5 ml of trivalent influenza vaccine, containing at least 15 microgram of hemagglutinin antigen per strain
  Interventions: Biological: seasonal influenza vaccine
- group 2 (Experimental): receives two-site intradermal dose of 0.1 ml each, containing at least 3 microgram of hemagglutinin antigen per strain per site
  Interventions: Biological: seasonal influenza vaccine
- group 3 (Experimental): receives two-site intradermal dose of 0.2 ml each, containing at least 6 microgram of hemagglutinin antigen per strain per site
  Interventions: Biological: seasonal influenza vaccine

INTERVENTIONS:
Biological: seasonal influenza vaccine — receives a single intramuscular dose of 0.5 ml of trivalent influenza vaccine, containing at least 15 microgram of hemagglutinin antigen per strain
  Other Names: influenza vaccine 2010 southern hemisphere; lot no 0700302A
  Arms: group 1
Biological: seasonal influenza vaccine — receives two-site intradermal dose of 0.1 ml each, containing at least 3 microgram of hemagglutinin antigen per strain per site and group
  Other Names: influenza vaccine 2010 southern hemisphere; lot no 0700302A
  Arms: group 2
Biological: seasonal influenza vaccine — receives two-site intradermal dose of 0.2 ml each, containing at least 6 microgram of hemagglutinin antigen per strain per site
  Other Names: influenza vaccine 2010 southern hemisphere; lot no 0700302A
  Arms: group 3

SUMMARY:
One-site dose sparing intradermal influenza vaccination in elderly had been studied but resulted in unsatisfactory outcomes. The investigators evaluate the safety and immunogenicity of the two-site intradermal injection of influenza vaccine containing all 6 and 12 micrograms of hemagglutinin antigen per strain (with 4/10th and 8/10th of a regular 15 microgram HA/strain intramuscular vaccine respectively) in elderly over 60 years of age. An influenza vaccine administered intramuscularly at the standard dose is used as the reference vaccine.

DETAILED DESCRIPTION:
The subjects would be randomly divided into three groups of 60 subjects each. Group1 receives a single intramuscular dose of 0.5 ml of trivalent influenza vaccine, containing at least 15 microgram of hemagglutinin antigen per strain, Group II receives two-site intradermal dose of 0.1 ml each, containing at least 3 microgram of hemagglutinin antigen per strain per site and group III receives two-site intradermal dose of 0.2 ml each, containing at least 6 microgram of hemagglutinin antigen per strain per site. Check for HA Antibody

ELIGIBILITY:
Inclusion Criteria:

* healthy male or female volunteer aged at least 60 years old
* willing to participate in this study

Exclusion Criteria:

* previous influenza vaccination within 6 months
* systemic ypersensitivity to egg or chicken proteins or any of the vaccine components
* history of a life-threatening reaction to the study vaccine or a vaccine containing the same constituents.
* ongoing acute febrile illness (oral temperature, ≥37.5 c )
* congenital or acquired immunodeficiency
* treatment with immunosuppressive or other immune- modifying drugs or cancer therapy within previous 6 months
* long-term treatment with systemic corticosteroids
* receipt of blood or blood-derived products in the previous 3 months
* history of thrombocytopenia or a bleeding disorder contraindicating for intramuscular vaccination.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2010-10; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
immunogenicity | 4 months
  evaluate the immunogenicity of the two-site intradermal influenza vaccination containing all 6 and 12 micrograms of hemagglutinin antigen per strain (with 4/10th and 8/10th of a regular 15 microgram HA/strain intramuscular vaccine respectively) in elderly over 60 years of age , as measured by the titer of hemagglutination inhibition (HAI) antibodies, in order to determine whether it would meet the guidelines of the European Committee for Proprietary Medicinal Products (CPMP) for the annual relicensure of influenza vaccines

SECONDARY OUTCOMES:
comparison of the immunogenicity | 4 months
  comparison of the immunogenicity of the two-site influenza vaccine administered intradermally as the above reduced dose with those of the reference influenza vaccine administered intramuscularly at the standard dose
safety | 4 months
  evaluate for number of participants with adverse effects:
  * systemic effects such as fever, headache, myalgia
  * local effects such as redness, swelling, induration and pain by giving diary card for each participant to record the data once daily for 1 week. (the investigators explain how to grade the redness (no/yes), swelling by measure, induration by measure, pain (no/yes))

CONTACTS AND LOCATIONS:
Overall Officials: Suda Sibunruang, MD, Principal Investigator — Queen Saovabha Memorial Institute
Locations (1):
- Queen Saovabha Memorial Institute, Bangkok, Thailand